CLINICAL TRIAL: NCT06437262
Title: Randomized Clinical Trial on the Immediate Antibacterial Effect and Substantivity of a Single Application of a New Chlorhexidine Gel on Oral Biofilm and Saliva
Brief Title: Antibacterial Effect and Substantivity of a New Chlorhexidine and Cymenol Gel on Oral Biofilm and Saliva
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Lacer S.A. (Industry)
Responsible Party: Principal Investigator, Inmaculada Tomás, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-CE161
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Healthy; Saliva; Biofilms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.20% CHX gel (Active Comparator): Participants underwent a single application of the 0.20% CHX gel. Samples were collected in basal conditions (i.e., before application) and at 5 minutes, 1 hour, 3 hours, 5 hours and 7 hours after application.
  Interventions: Drug: 0.20% CHX gel on saliva; Drug: 0.20% CHX gel on oral biofilm
- 0.20% CHX and Cymenol gel (Experimental): Participants underwent a single application of the 0.20% CHX + Cymenol gel. Samples were collected in basal conditions (i.e., before application) and at 5 minutes, 1 hour, 3 hours, 5 hours and 7 hours after application.
  Interventions: Drug: 0.20% CHX and Cymenol gel on saliva; Drug: 0.20% CHX and Cymenol gel on oral biofilm

INTERVENTIONS:
Drug: 0.20% CHX gel on saliva — In vivo application of a gel on the vestibular and palatal/lingual gingival mucosa of both arches at minute 0 for posterior saliva collection at different time-points.
  Arms: 0.20% CHX gel
Drug: 0.20% CHX and Cymenol gel on saliva — In vivo application of a gel on the vestibular and palatal/lingual gingival mucosa of both arches at minute 0 for posterior saliva collection at different time-points.
  Arms: 0.20% CHX and Cymenol gel
Drug: 0.20% CHX gel on oral biofilm — Ex vivo application of a gel on the glass disks of the removable intraoral appliance at minute 0 for subsequent one-by-one disk removal from the device at different time-points.
  Arms: 0.20% CHX gel
Drug: 0.20% CHX and Cymenol gel on oral biofilm — Ex vivo application of a gel on the glass disks of the removable intraoral appliance at minute 0 for subsequent one-by-one disk removal from the device at different time-points.
  Arms: 0.20% CHX and Cymenol gel

SUMMARY:
The objective of this project was to compare the immediate antimicrobial effect and in situ substantivity of a new 0.20% chlorhexidine (CHX) gel and cymenol with the current CHX gel formulation on dental plaque biofilm and salivary flora up to 7 hours after a single application.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy volunteers
* Age between 20-45 years
* Presence of minimum 24 permanent teeth
* No evidence of gingivitis or periodontitis (CPITN= 0)
* No presence of untreated caries at the start of the study

Exclusion Criteria:

* Smoker or ex-smoker
* Presence of dental protheses or orthodontic appliances
* Antibiotic treatment and/or routine use of oral antiseptics in the previous three months
* Presence of any systemic disease that could alter saliva production or composition

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Intragel bacterial viability: baseline vs 5 minutes | Baseline, 5 minutes
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) with either 0.20% CHX gel or 0.20% CHX and cymenol gel: baseline vs 5 minutes
Intragel bacterial viability: baseline vs 1 hour | Baseline, 1 hour
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) with either 0.20% CHX gel or 0.20% CHX and cymenol gel: baseline vs 1 hour
Intragel bacterial viability: baseline vs 3 hours | Baseline, 3 hours
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) with either 0.20% CHX gel or 0.20% CHX and cymenol gel: baseline vs 3 hours
Intragel bacterial viability: baseline vs 5 hours | Baseline, 5 hours
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) with either 0.20% CHX gel or 0.20% CHX and cymenol gel: baseline vs 5 hours
Intragel bacterial viability: baseline vs 7 hours | Baseline, 7 hours
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) with either 0.20% CHX gel or 0.20% CHX and cymenol gel: baseline vs 7 hours
Intragel bacterial viability: 5 minutes vs 1 hour | 5 minutes, 1 hour
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) with either 0.20% CHX gel or 0.20% CHX and cymenol gel: 5 minutes vs 1 hour
Intragel bacterial viability: 5 minutes vs 3 hours | 5 minutes, 3 hours
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) with either 0.20% CHX gel or 0.20% CHX and cymenol gel: 5 minutes vs 3 hours
Intragel bacterial viability: 5 minutes vs 5 hours | 5 minutes, 5 hours
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) with either 0.20% CHX gel or 0.20% CHX and cymenol gel: 5 minutes vs 5 hours
Intragel bacterial viability: 5 minutes vs 7 hours | 5 minutes, 7 hours
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) with either 0.20% CHX gel or 0.20% CHX and cymenol gel: 5 minutes vs 7 hours
Intergel bacterial viability at baseline: 0.20% CHX gel vs 0.20% CHX and cymenol gel | Baseline
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) at baseline: 0.20% CHX gel vs 0.20% CHX and cymenol gel.
Intergel bacterial viability after 5 min: 0.20% CHX gel vs 0.20% CHX and cymenol gel | 5 minutes
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) after 5 minutes: 0.20% CHX gel vs 0.20% CHX and cymenol gel.
Intergel bacterial viability after 1 hour: 0.20% CHX gel vs 0.20% CHX and cymenol gel | 1 hour
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) after 1 hour: 0.20% CHX gel vs 0.20% CHX and cymenol gel.
Intergel bacterial viability after 3 hours: 0.20% CHX gel vs 0.20% CHX and cymenol gel | 3 hours
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) after 3 hours: 0.20% CHX gel vs 0.20% CHX and cymenol gel.
Intergel bacterial viability after 5 hours: 0.20% CHX gel vs 0.20% CHX and cymenol gel | 5 hours
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) after 5 hours: 0.20% CHX gel vs 0.20% CHX and cymenol gel.
Intergel bacterial viability after 7 hours: 0.20% CHX gel vs 0.20% CHX and cymenol gel | 7 hours
  Percentage of bacterial viability (Ratio of viable bacteria to total bacteria -viable + non-viable- multiplied by 100) after 7 hours: 0.20% CHX gel vs 0.20% CHX and cymenol gel.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Tomás, Prof, Principal Investigator — University of Santiago de Compostela, Spain
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No